CLINICAL TRIAL: NCT03288623
Title: The Effects of Dark Chocolate Implementation in the Reduction of Oxidative Stress and Improvement of Vascular Function and Physical Performance in Elite Athletes
Brief Title: The Effects of Dark Chocolate Implementation in Elite Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Elena Cavarretta, MD, PhD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE 4662
Record Dates: First submitted 2017-09-14; First posted 2017-09-20 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Oxidative Stress; Athletes Heart; Physical Activity
MeSH Terms: conditions — Motor Activity | interventions — Chocolate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dark Chocolate (Experimental): Dark chocolate (85% cocoa) 40 mg per day for 30 days
  Interventions: Dietary Supplement: Dark Chocolate (85% cocoa)
- White/Milk Chocolate (Placebo Comparator): White chocolate or Milk chocolate administration in tablet (<35% cocoa) per day for 30 days
  Interventions: Dietary Supplement: White/Milk chocolate (<35% cocoa)

INTERVENTIONS:
Dietary Supplement: Dark Chocolate (85% cocoa) — Dark chocolate (85% cocoa) in tablet
  Arms: Dark Chocolate
Dietary Supplement: White/Milk chocolate (<35% cocoa) — white or milk chocolate (<35% cocoa) in tablet
  Arms: White/Milk Chocolate

SUMMARY:
Dark chocolate (DC) is rich in epicatechin which augments nitric oxide (NO) production through endothelium-dependent influences. The increased bioavailability and activity of NO have been demonstrated to statistically increase flow-mediated dilation in healthy subjects and in hypertensive patients. DC supplementation has been hailed for its positive effects on cardiovascular health and it has been proposed as a booster of physical performance in athletes, however the mechanisms by which DC improves oxidative stress, vascular function and athletic performance are not fully understood. The investigators designed a human study assessing how DC improves NO bioavailability and activity in elite athletes. Twenty-four elite soccer players (aged 18-35 years old, all males) are divided in 2 groups and randomly assigned to receive DC (85% cocoa), 40g per day or white/milk chocolate (<35% cocoa) for 30 days. The primary outcome measure is the evaluation of Soluble NOX2-derived peptide (sNOX2-dp), a direct marker of NADPH oxidase activation. The secondary outcome measures are other markers of oxidative stress, as the soluble P-selectin (sPs), Vitamin E, soluble CD40 Ligand (sCD40L), a marker of in vivo platelet activation and flow-mediated dilation assessed by vascular ultrasound. All parameters are assessed at baseline and after 30 days in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Elite male athletes volunteers, aged between 18 and 35 years

Exclusion Criteria:

* they suffer from an allergy to cocoa or any of the ingredients contained within either of the chocolate bars
* they have a low platelet count (< 170 x 10E09/ L)
* they are taking aspirin or aspirin-containing drugs, other anti-inflammatory drugs, or any drugs or herbal medicines known to alter platelet function or the haemostatic system in general (without a minimum washout period of one month)
* they are taking fish oils or evening primrose oil, or fat soluble vitamin supplements within the last 4 weeks
* they have unsuitable veins for blood sampling and/ or cannulation
* they have a BMI below 18 or above 35 kg/ sqm
* they are taking any medicine known to affect lipid and/or glucose metabolism
* they are suffering from alcohol or any other substance abuse or are having eating disorders
* they have any known clinical signs of diabetes, hypertension, renal, hepatic, hematological disease, gastrointestinal disorders, endocrine disorders, coronary heart disease, infection or cance

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Soluble NOX2-derived peptides (sNOX2-dp) | 30 days
  a marker of nicotinamide adenine dinucleotide phosphateoxidase activation, was detected in serum by ELISA. The peptide was recognised by the speciﬁc monoclonal antibody against the amino-acidic sequence (224-268) of the extra membrane portion of NOX2. Values were expressed as pg/mL; intra-assay and inter-assay coefﬁcient of variation is 5%

SECONDARY OUTCOMES:
soluble P-selectin (sPs) | 30 days
  soluble P-selectin levels, a marker of in-vivo platelet activation, will be measured on citrated platelet poor plasma samples by enzyme immunoassay
soluble CD40 Ligands (sCD40L) | 30 days
  soluble CD40 Ligand, a marker of in vivo platelet activation, will be measured using a commercially available method by Luminex Technology according to the manufacturer's instructions (Milliplex Map Kit Millipore, Darmstadt, Germany) in platelet components
Hydrogen Peroxide (H2O2) | 30 days
  Hydrogen peroxide (H2O2) is produced by inflammatory and vascular cells. Extracellular H2O2 is detected using incubation with Amplex Red (10 μM) and horseradish peroxidase (0.2 U/mL) for 60 min at 37 °C in Krebs-Ringer's phosphate glucose buffer (in mM: 145 NaCl, 5.7 sodium phosphate, 4.86 KCl, 0.54 CaCl2, 1.22 MgSO4, and 5.5 glucose) protected from light. Fluorescence is detected at 590 nm using an excitation of 530 nm every 5 min for 60 min. H2O2 is expressed as fluorescence per minute.
flow-mediated dilation (FMD) | 30 days
  Evaluation of brachial artery FMD was performed at 60 seconds (FMD60s) and 120 seconds (FMD120s) postischemic stress by vascular ultrasound. Early FMD was defined as peak FMD60s and delayed FMD as peak FMD120s.
Vitamin E (α-tocopherol, αT) | 30 days
  Serum samples will be supplemented with tocopheryl acetate (internal standard), deproteinized by the addition of ethanol, and extracted with hexane. Phase separation is achieved by centrifugation. The collected upper phase is evaporated and analysed using an Agilent 1200 Infinity series high-performance liquid chromatography system equipped with an Eclipse Plus C18 column (4.6 × 100 mm). Serum levels will be given as the ratio (μmol/mmol) between serum α-tocopherol concentration (μmol/L) and serum total cholesterol concentration (mmol/L), which better express the circulating levels of vitamin E.
Serum isoprostane (8-iso-PGF2a-III) | 30 days
  Serum isoprostane (8-iso-PGF2a-III) is measured by the enzyme immunoassay method (DRG International). The values are expressed as pmol/l.

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Frati, MD, Study Director — University of Roma La Sapienza
Locations (1):
- Sapienza University of Rome, Policlinico Umberto I, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual participant data for all primary and secondary outcome measures will be made available

REFERENCES:
- [Result] Cavarretta E, Peruzzi M, Del Vescovo R, Di Pilla F, Gobbi G, Serdoz A, Ferrara R, Schirone L, Sciarretta S, Nocella C, De Falco E, Schiavon S, Biondi-Zoccai G, Frati G, Carnevale R. Dark Chocolate Intake Positively Modulates Redox Status and Markers of Muscular Damage in Elite Football Athletes: A Randomized Controlled Study. Oxid Med Cell Longev. 2018 Nov 21;2018:4061901. doi: 10.1155/2018/4061901. eCollection 2018. PMID 30584461